CLINICAL TRIAL: NCT02244931
Title: Comparison of Three Assisting Devices to Power Manual Wheelchairs in Patients With Spinal Cord Injury : Assessment of Biomechanical, Physiological and Functional Properties.
Brief Title: Comparison of Three Different Assisting Devices to Power Manual Wheelchairs in Patients With Spinal Cord Injury
Acronym: PAPAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2011-A00151-40
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injuries, paraplegic, manual wheelchairs, assisting propelling device
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1: Performance evaluation on ergometer (Experimental): The 3 devices are experimented in random order to compare them on performance using an ergometer wheelchair:
  * Servomatic™ assisting device
  * E.Motion© assisting device
  * Standard manual Wheelchair
  Interventions: Device: Servomatic™ assisting device; Device: E.Motion© assisting device; Device: Standard manual Wheelchair
- Phase 2: Comparison of maneuverability (Experimental): The 3 devices are experimented in random order to compare them on maneuverability:
  * Servomatic™ assisting device
  * E.Motion© assisting device
  * Standard manual Wheelchair
  Interventions: Device: Servomatic™ assisting device; Device: E.Motion© assisting device; Device: Standard manual Wheelchair
- Phase 3: Comparison of the autonomy (Experimental): The 3 devices are experimented in random order to compare them on the autonomy they afford to patients:
  * Servomatic™ assisting device
  * E.Motion© assisting device
  * Standard manual Wheelchair
  Interventions: Device: Servomatic™ assisting device; Device: E.Motion© assisting device; Device: Standard manual Wheelchair

INTERVENTIONS:
Device: Servomatic™ assisting device — Servomatic™ is an hand controlled motorized device assisting to propel the wheelchair .
Device: E.Motion© assisting device — E.Motion© is an hand controlled motorized device assisting to propel the wheelchair .
Device: Standard manual Wheelchair — Standard manual Wheelchair

SUMMARY:
The purpose of this study is to compare three assisting devices to propel personal wheelchairs (Servomatic A©, Servomatic B© and E.Motion©) to the standard personal manual wheelchair in patients with spinal cord injury.

DETAILED DESCRIPTION:
The objective of the study is to compare three assisting devices to propel personal wheelchairs (Servomatic A©, Servomatic B© and E.Motion©) to the standard personal manual wheelchair in patients with spinal cord injury.

The study consists of three distinct and independent phases:

* Phase 1: Performance evaluation on wheelchair ergometer in order to compare the energy expenditure and kinetic characteristics in comparable situations with regard to speed and workload imposed to the wheelchair-patient couple.
* Phase 2: Comparison of maneuverability and ease of crossing usual obstacles in outdoor and indoor paths with standardised obstacles. Trajectories are to be recorded in order to allow analysis by independent experts.
* Phase 3: Comparison of the autonomy of patients afforded by the devices by comparing the patient's ability to transfer from wheelchair to car seat and from car seat to wheelchair, as well as ease of wheelchair packing in car, in the context of a standard city transport involving a car and the wheelchair.

The three phases are to be performed using the standard manual wheelchair and the three assisting devices in a randomized order.

Three different groups of patients are included in the three phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 70 years
* Spinal cord injury C5-C8, paraplegic D1-D11, and D11 paraplegic below only for phases 1 and 2 phase 1 and 2
* Spinal cord injury D1 and above only for phase 3
* Having given free and informed consent
* Negative pregnancy test for women of childbearing age

Exclusion Criteria:

* No affiliation to a social security scheme
* Refusal to participate in the clinical trial
* Patient under guardianship
* Major cognitive disorders
* bedsores
* Functional abnormality of the shoulder
* History of cardiovascular disease
* ECG to suspect coronary insufficiency
* Pregnant patients without effective treatment or contraceptive
* Acute complication or systemic organ

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Phase 1: physiological parameters : Oxygen consumption. | 3 hours
Phase 2: Ease of crossing obstacles assessed by patients with a Visual Analog Scale | 3 hours
Phase 3: Time necessary to transfer from wheelchair to car and from car to wheelchair. | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nadine NP PELLEGRINI, MD, Principal Investigator — Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, 92380 Garches, France
Locations (1):
- Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, Garches, France

REFERENCES:
- [Derived] Guillon B, Van-Hecke G, Iddir J, Pellegrini N, Beghoul N, Vaugier I, Figere M, Pradon D, Lofaso F. Evaluation of 3 pushrim-activated power-assisted wheelchairs in patients with spinal cord injury. Arch Phys Med Rehabil. 2015 May;96(5):894-904. doi: 10.1016/j.apmr.2015.01.009. Epub 2015 Jan 22. PMID 25620717